CLINICAL TRIAL: NCT01086735
Title: Suicide Gene Therapy for Donor Lymphocytes Infusion After Allogeneic Hematopoietic Stem Cell Transplantation: a Phase I/II Clinical Study
Brief Title: Suicide Gene Therapy for Donor Lymphocytes Infusion After Allogeneic Hematopoietic Stem Cell Transplantation
Acronym: ILD-TK01
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Paris 12 Val de Marne University (Other); Pierre and Marie Curie University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P010506
Record Dates: First submitted 2010-03-12; First posted 2010-03-15 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Hematological Malignancy
Keywords: hematological malignancy; allogeneic hematopoietic stem cell transplantation; donor lymphocyte infusion; antitumor immunotherapy; graft-versus-tumor effect; gene therapy; relapse; adult
MeSH Terms: conditions — Hematologic Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- donor lymphocyte infusion (Experimental): Donor T-cell transduction
  Interventions: Biological: donor lymphocyte infusion

INTERVENTIONS:
Biological: donor lymphocyte infusion — Donor T-cell transduction

SUMMARY:
The main complications of allogeneic hematopoietic stem cell transplantation (HSCT) include graft-versus-host disease (GVHD) and poor immune reconstitution leading to severe infections and leukemia relapse. Mature donor T-cells present in the transplant facilitate T-cell reconstitution but also induce GVHD, which itself impairs immune reconstitution. We have developed a strategy of alloreactive T-cell depletion, using T-cells expressing the Herpes simplex thymidine kinase (TK) suicide gene combined with a ganciclovir (GCV) treatment. This system permits the selective elimination of dividing TK+ T-cells in vivo. To test this hypothesis in preclinical settings, we have previously developed several experimental models of GVHD using TK+ T-cells in mice. The demonstration that a preventive treatment with GCV administered close to the time of HSCT could control GVHD brought the proof of concept. We now propose a clinical trial to test whether donor lymphocytes infusion (DLI) using TK-transduced cells permits to induce a graft-versus-tumor (GVT) effect for treatment of relapse after HSCT, while GVHD can be controlled by GCV treatment.

DETAILED DESCRIPTION:
DLI-TK is administered either after failure of 1 or several previous standard (std-) DLI of, defined after a minimal follow-up of 2 months after the last injection. To prepare DLI-TK, donor T-cells are transduced with a retroviral vector encoding TK. Transduced cells are selected using a CliniMACS device (MYLTENYI). In case of previous std-DLI received, the DLI-TK cell dose is adjusted to be below or equal to the maximal cell dose previously received in std-DLI. No comparison is planned in the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Hematological malignancy.
* Previous allogeneic hematopoietic stem cell transplantation.
* Relapse diagnosed at the molecular, cytogenetic, or cytological level.
* Failure of a previous stdILD or inclusion in first intention without previous stdDLI.
* Age > 18 years and < 70 years at the time of inclusion. For patients between 15 and 18 years of age, a case-per case inclusion will be studied.
* Performance status considered on the score Eastern Cooperative Oncology Group (ECOG) < 2.
* Life expectation 1-month-old superior.
* Signed written informed consent.
* Negative human chorionic gonadotropin (HCG) in the 7 days preceding the inclusion for women in age of procreation.
* Membership of the French national insurance.

Exclusion Criteria:

* Grade >II acute GVHD or chronic extensive GVHD at the time of inclusion.
* Patient receiving an immunosuppressive treatment for GVHD treatment at the time of inclusion.
* Dysfunction of liver (alanine aminotransferase / aspartate transaminase (ALAT/ASAT) > 5 N, or bilirubin > 50 µM), or of the renal function (creatinine clearance < 30 ml / min).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-02; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Incidence of "severe" GHVD (acute grade >II or chronic extensive) following DLI-TK and treatment with GCV | during the 12 months of follow-up
  Incidence of "severe" GHVD (acute grade >II or chronic extensive) following DLI-TK and treatment with GCV

SECONDARY OUTCOMES:
The incidence of GVHD of any grade after DLI-TK | during the 12 months of follow-up
  The incidence of GVHD of any grade after DLI-TK
The anti-tumoral efficiency of DLI-TK to treat the relapse of the hematological malignancy | during the 12 months of follow-up
  The anti-tumoral efficiency of DLI-TK to treat the relapse of the hematological malignancy
The survival and the survival without disease after DLI-TK | during the 12 months of follow-up
  The survival and the survival without disease after DLI-TK

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Maury, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Groupe Hospitalier Albert Chenevier-Henri Mondor, Créteil, France